CLINICAL TRIAL: NCT05928234
Title: A Longterm Follow-up and Comparison of Morbidity and Heart Health Between Patients With Pulmonary Atresia With Intact Ventricular Septum and Uni- or Biventricular Circulation
Brief Title: A Comparison of Morbidity Between Patients With Pulmonary Atresia With Intact Ventricular Septum and Uni- or Biventricular Circulation
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Stina Manhem, MD, Vastra Gotaland Region
Other Study IDs: PA-IVS, 2023
Record Dates: First submitted 2023-06-04; First posted 2023-07-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Atresia With Intact Ventricular Septum
MeSH Terms: conditions — Pulmonary Atresia with Intact Ventricular Septum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biventricular circulation: Research subjects with PA-IVS who have biventricular circulation
- Univentricular circulation: Research subjects with PA-IVS who have univentricular circulation

SUMMARY:
The goal of this observational study is to compare patients with pulmonary atresia with intact ventricular septum (PA-IVS) with univentricular circulation to patients with the same heart defect but that has a biventricular circulation in regards to mortality, quality of life, comorbidity, cardiac function, and work capacity. The main questions the study aims to answer are:

• Do mortality, quality of life, comorbidity, cardiac function, and work capacity differ between patients with PA-IVS who have univentricular and biventricular circulation?

Participants will be asked to answer a Quality of Life questionnaire. The investigators will also inquire with a sample size of the research subjects (based on place of residence) about their participation in a series of examinations (ergo-spirometry to assess work capacity, transthoracic echocardiogram, magnetic resonance of the heart and blood sampling to assess cardiac function and cardiac health).

ELIGIBILITY:
Inclusion Criteria:

* Individuals born with pulmonary atresia with intact ventricular septum (PA-IVS) who are 15 years or older at the start of the study.
* Regarding the mortality variable, research subjects who have died after the age of 15 years old will be included.

Exclusion Criteria:

Individuals born with pulmonary atresia with intact ventricular septum who are younger than 15 years old at the start of the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all individuals with PA-IVS who have been registered in Swedcon (a national register for patients with congenital heart defects) or in the National Patient Register and Cause of Death Register since 1980 and meet other inclusion criteria, including age.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Difference in comorbidity between the two groups | September 2024
  Difference in myocardial infarction, heart failure, arrhythmia, stroke, malignancy, autoimmune diseases, infections, atopy, certain liver diseases, and protein-losing enteropathy between the two groups

SECONDARY OUTCOMES:
Difference in quality of life between the two groups | September 2024
  A validated quality of life questionnaire (PROMIS Scale v1.2-Global Health) will be sent to all the research subjects and the answers will be compared between the two groups. The questionnaire consists of a ten-item patient reported measure of physical, mental and social health. Each statement is answered on a scale from 1-5, higher scores mean better outcome.
Difference in physical capacity between the two groups | September 2024
  Ergospirometry, outcome variables: exercise test (exercise capacity measured in watt and over time, counted in minutes), oxygen saturation (measured in percent), blood pressure (measured in millimetre of mercury)
Difference in cardiac capacity between the two groups | September 2024
  Transthoracic echocardiogram
Difference in general health, linked to cardiac health, between the two groups | September 2024
  The following blood tests will be analysed: N-terminal pro-brain natriuretic peptide (a marker for heart failure), Alanine aminotransferase (a liver enzyme), Aspartate aminotransferase (a liver enzyme), Creatinine (a waste product from muscle metabolism, used to assess kidney function), Sodium (an electrolyte), Potassium (an electrolyte), Hemoglobin (a protein in red blood cells that carries oxygen), White blood cell count (Leukocyte count), Platelet count (Thrombocyte count), Albumin: A protein produced by the liver that helps maintain fluid balance in the body, TREC (T-receptor excision circles): A marker used to assess immune function, specifically the production of new T cells, Expanded lymphocyte typing (a comprehensive examination of lymphocyte subtypes)
Difference in mortality between the groups | September 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Heart Center, Queen Silvia's Children's hospital, Gothenburg, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT05928234/Prot_SAP_000.pdf